CLINICAL TRIAL: NCT03318172
Title: High-Density Spinal Cord Stimulation for the Treatment of Chronic Intractable Pain Patients: A Prospective Multicenter Randomized Controlled, Double-blind, Crossover Exploratory Study With 6-m Open Follow-up
Brief Title: High-Density Spinal Cord Stimulation for the Treatment of Chronic Intractable Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruting of patients
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Clinical Associate Professor, Seoul National University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1703-133-841
Record Dates: First submitted 2017-10-16; First posted 2017-10-23 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pain, Intractable
Keywords: Spinal Cord Stimulation; High Density Stimulation
MeSH Terms: conditions — Pain, Intractable

STUDY DESIGN:
Intervention Model Description: V1 SCS trial for 6 days (3d conventional + 3d HD stimulation).
  V2 Enrolled if positive response (≥50% pain reduction) in one of the two modes during V1 + informed consent and randomization + blinding
  * Group C Conventional mode (2 weeks) + HD mode (2 weeks)
  * Groups H HD mode (2 weeks) + conventional mode (2 weeks)
  V3 After 2 weeks (+3d allowed) from V2. Cross-over performed by the MedTronics person in charge of adjusting the SCS mode. Mode-related information will not be shared with other researchers
  V4 (unblinding) 2 weeks from V3 (+3d allowed). Patients will be questioned about the more effective mode (primary endpoint). The SCS will be programmed accordingly
  V5 (follow-up 1) 4 weeks after V4 (±5d). Short-term assessment of effectiveness and safety
  V6 (follow-up 2) 12 weeks after V4 (±5d). Middle-term assessment of effectiveness and safety
  V7 (follow-up 3) 24 weeks after V4 (±5d). Long-term assessment of effectiveness and safety
Who Masked: Participant, Care Provider, Investigator
Masking Description: The day of the SCS implantation (RestoreSensor Surescan MRI Neurostimulator, Medtronic ©) the patients are randomized based on a random number assigned from www.randomization.com. The random number table is sent to the MedTronic representative in charge of the SCS mode control by the operating nurse who has no information about the study protocol. At this time, implantation practitioners and other research participants don't know which group is assigned first. Subjects with SCS implantation will be assigned 1:1 to either group C (conventional stimulation) or H (High-Density stimulation) to find an effective mode of pain relief.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group C spinal cord stimulator (Experimental): Spinal cord stimulator (SCS) implantation with conventional stimulation mode therapy during 2 weeks followed by 2 weeks with high-density stimulation mode therapy.
  Interventions: Device: Spinal Cord Stimulator
- Group H spinal cord stimulator (Active Comparator): Spinal cord stimulator (SCS) implantation with high-density stimulation mode therapy during 2 weeks followed by 2 weeks with conventional stimulation mode therapy.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — Implantation of spinal cord stimulator in patients included in the study and divided in conventional and high density stimulation groups
  Other Names: Conventional stimulation mode; High density stimulation mode

SUMMARY:
The purpose of this study is to explore which mode is effective in the management of intractable chronic pain, the high-density stimulation or the conventional stimulation, in patients who undergo SCS implantation after successful pre-implantation SCS trial.

DETAILED DESCRIPTION:
Since its introduction in 1967 (1), spinal cord stimulation (SCS) has become a well-established modality for the treatment of chronic neuropathic back and leg pain, including postlaminectomy syndrome, complex regional pain syndrome, ext. (2-5) The mechanism of action remains poorly understood but is thought to involve a combination of local neural inhibition, excitation of nearby axons, changes in neurotransmitter physiology, and jamming of pathological network activity by masking intrinsic patterns of neural activity (6). It is generally agreed that a sensory percept (paresthesia) covering the region of pain is required in order to achieve maximal effectiveness (3,7), and as a result, conventional SCS settings typically consist of intermediate frequencies (40-60 Hz), relatively long pulse width (300-500 μsec), and amplitude high enough to induce a sensory percept in the distribution of the patient's pain (2,3,5). However, paresthesia can produce some degree of discomfort, particularly with changes in position and variability of activities (8). Consequently, sometimes there is a trade-off between pain relief and paresthesia discomfort, and the clinical benefits can be offset by the side-effects of the stimulation. Recent studies have attempted to deliver energy to the spinal cord below the threshold for paresthesia ("paresthesia-free" stimulation), with variable degrees of success in the control of neuropathic pain. For example, De Ridder et al. described "burst" stimulation (trains of five pulses) in 12 patients, resulting in paresthesia-free pain relief that was superior to conventional settings (9). In a multicenter prospective study, Al-Kaisy et al. evaluated 10 kHz SCS (HFSCS) delivered below the sensory threshold and documented a long-term reduction in the mean intensity of chronic back pain (10). However, a randomized, double-blind, placebo-controlled crossover study comparing 5 kHz high-frequency subthreshold stimulation to placebo found no significant difference between the two modalities, with a tendency for better results during the first treatment administered, which suggests a strong placebo effect (11). Another randomized controlled, double-blinded, crossover study showed that subthreshold stimulation had significantly lower pain relief than the conventional, supra-threshold SCS (12). Notably, both studies included participants treated with conventional stimulation parameters and did not perform a "trial" to confirm that the study population would, in fact, demonstrate a response to subthreshold stimulation. Most systematic studies of paresthesia-free stimulation employed a high rate of energy delivery (high-density [HD] stimulation) that either required the development of specialized hardware (9,10) or modification of existing systems to allow parameters outside of normal clinical use (11). However, it is possible that rechargeable stimulators currently in widespread use may be able to deliver sufficient energy to accomplish pain relief without paresthesia in appropriately selected patients. Additionally, response to subthreshold stimulation might be heterogeneous in unpredictable ways, which implies that there might be a subset of patients who respond to the therapy better than others.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic intractable pain who meets the Korean SCS Reimbursement Guideline as follows:

   (Korea SCS Reimbursement Guideline)
   1. An ineffective patient with sustainable severe intractable pain (VAS or NRS pain score over 7 grade) who has been treated by a conservative therapy (medication and nerve block, etc.) for 6 months. cf.) CRPS is available after the conservative therapy for 3 months
   2. An ineffective cancer pain patient with over 1-year life expectancy and VAS (or NRS pain score) over 7 grade who takes active pain treatment for 6 months such as medication, nerve block, epidural morphine injection, etc.
2. Age > 18
3. Patients who have been informed of the study procedures and has given written informed consent.
4. Patients who are willing to comply with study protocol including attending the study visits

Exclusion Criteria:

1. Expected inability of patients to receive or properly operate the SCS system
2. Active malignancy
3. Addiction to any of the following drugs, alcohol, and/or medication
4. Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
5. Local infection or other skin disorder at site of incision
6. Pregnancy
7. Other implanted active medical device
8. Life expectancy < 1 year
9. Coagulation deficiency (Platelet count < 100,000, PT INR > 1.4)
10. Immune deficiency (HIV positive, immunosuppressive, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Percentage of high density SCS mode selected by participants | Four weeks after randomization
  Patients will be questioned about the more effective mode of pain relief between conventional and high density stimulation.

SECONDARY OUTCOMES:
Difference of pain intensity between the baseline screening and the evaluation at each visit | Six month from baseline screening
  Pain intensity will be evaluated using NRS (0-10) pain score
Change of pain characteristics between the baseline screening and the evaluation at each visit | Six month from baseline screening
  The pain characteristics will be evaluated using PainDETECT
The ability in daily living | Screening and follow up at 1 month, 3 months and 6 months
  Measured by the Korean version of the Instrumental Activities of Daily Living (K-IADL) scale. The IADL require complex thinking skills, including organizational skills and they measure the ability of the person to live independently without the assistance of another person.
  The IADL scale includes 8 categories labeled from A to H (A. Ability to Use Telephone, B. Shopping, C. Food preparation, D. Housekeeping, E. Laundry, F. Mode of transportation, G. Responsibility for Own Medication and H. Ability to Handle Finances). For each category, the patient should mark the description that resembles the highest functional level (either 0 or 1). A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
The current pain intensity and interference status | Screening and follow up at 1 month, 3 months and 6 months
  The Brief Pain Inventory Short-Form (BPI-SF) scale measures the pain intensity (severity) and the impact of pain on functioning (interference). Includes a screening question about the pain on the day, pain drawing diagrams, four items about pain intensity (worst pain, least pain, average pain, pain right now), two items on pain relief treatment or medication, and one item on pain interference, with seven sub-items (general activity, mood, walking ability, normal walk, relations with other people, sleep, and enjoyment of life). Each item for pain severity is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score (0 to 40). The seven subitems of pain interference are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score (0 to 70). The first item, pain drawing diagrams and the items on pain relief treatment or medication do not contribute to the scoring.
Subjective sleep quality | Screening and follow up at 1 month, 3 months and 6 months
  The difference of Insomnia Severity Index (ISI) between the baseline screening and the evaluation at 1 month, 3 months and 6 months follow up visits
Oswestry Disability Index | Screening and follow up at 1 month, 3 months and 6 months
  The difference of Oswestry Disability Index between the baseline screening and the evaluation at 1 month, 3 months and 6 months follow up visits
Beck Depression Inventory | Screening and follow up at 1 month, 3 months and 6 months
  The difference of Beck Depression Inventory between the baseline screening and the evaluation at 1 month, 3 months and 6 months follow up visits
Pain Catastrophizing scale | Screening and follow up at 1 month, 3 months and 6 months
  Pain catastrophizing is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event. The Pain Catastrophizing Scale (PCS) is a 13-item instrument derived from definitions of catastrophizing described in the literature. The PCS ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales from (0) not at all and (4) all the time. The PCS total score is computed by summing responses to all 13 items, total scores range from 0 - 52. The PCS subscales are computed as follows:
  Rumination: Sum of items 8, 9, 10, 11 Magnification: Sum of items 6, 7, 13 Helplessness: Sum of items 1, 2, 3, 4, 5, 12 Total score <30= Negative and ≥30= Positive for catastrophizing
The Connor-Davidson Resilience Scale (CD-RISC) | Screening and follow up at 1 month, 3 months and 6 months
  Resilience embodies the personal qualities that enable one to thrive in the face of adversity. The Connor-Davidson Resilience Scale (CD-RISC) contains 25 items, all of which carry a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all the time (4). The scale is rated based on how the subject has felt over the past month.
  The total score ranges from 0-100, with higher scores reflecting greater resilience.
Patient Global Impression of Change (PGIC) | Follow up visits 1 month, 3 months and 6 months
  The overall change in patient's pain for 6 months after the study unblinding, during the follow up visits
Clinical Global Impressions-Improvement (CGI-I) | Follow up visits 1 month, 3 months and 6 months
  The overall change in patient's improvement for 6 months after the study unblinding, during the follow up visits
Patient's satisfaction with the stimulation mode | Follow up visits 1 month, 3 months and 6 months
  The difference in the patient's satisfaction evaluated during the follow-up visits using a 5-point Likert scale (5: very satisfied, 4: somewhat satisfied, 3: Dissatisfied, 1: very unsatisfied)
Any change of pain medication | Six month from baseline screening
  The difference between the baseline screening and the evaluation at each visit
Pain area coverage by the SCS | Crossover and follow-up visits 1 month, 3 months and 6 months
  The difference between crossover and follow-up visits (total of 5 times evaluation) by the patient drawing the area of pain coverage. The ideal treatment with SCS will be a total coverage of the pain area, however, sometimes the covered area does not perfectly match with the stimulated area (less or more area). Therefore, a simple drawing of a human body will be presented to the patients who will draw the area of pain and then the coverage of the SCS to compare and analyze the changes throughout the study.
Paresthesia threshold | Randomization, crossover and follow-up visits 1 month, 3 months and 6 months
  The difference between the randomization, crossover and follow-up visits (total of 6 evaluation) by asking patient to indicate the threshold at which he or she experiences paresthesia. The SCS transmitter allows several intensity levels which are tested before setting the SCS mode. Usually, the intensity level is tested from lowest and slowly increased until the patient experience paresthesia. Paresthesia threshold is different from patient to patient and it might change along time. Therefore, the intensity level marked by the SCS transmitter where the patient experienced the paresthesia will be recorded to evaluate the changes during the study period.
Change in the overall SCS stimulation parameters | From week 1 (randomization) to 6 months follow-up visit
  SCS stimulation parameters (active electrodes, frequency, pulse duration, amplitude and battery consumption) each visit after implantation. All parameters of SCS will be recorded in the same item as they are measured based on the SCS transmitter records and reflect the overall SCS status.
Battery efficiency of the neuro-stimulator | Follow up visits 1 month, 3 months and 6 months
  The battery usage will be measured by frequencies to recharge the battery during the follow-up visits.
Adaptive Stim use | Follow up visits 1 month, 3 months and 6 months
  Acquire information on activity from the internal diary; amount of times that patients need to fit the ideal parameters themselves) during the follow-up visits
Measurement of adverse events | Six month from baseline screening
  Any related adverse events throughout the whole study period (e.g. infection, hematoma, seroma, lead breakage, lead migration, SCS removal, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Jee Y Moon, PhD, Principal Investigator — Clinical Associate Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shealy CN, Mortimer JT, Reswick JB. Electrical inhibition of pain by stimulation of the dorsal columns: preliminary clinical report. Anesth Analg. 1967 Jul-Aug;46(4):489-91. No abstract available. PMID 4952225
- [Background] North RB, Kidd DH, Farrokhi F, Piantadosi SA. Spinal cord stimulation versus repeated lumbosacral spine surgery for chronic pain: a randomized, controlled trial. Neurosurgery. 2005;56(1):98-106; discussion 106-7. doi: 10.1227/01.neu.0000144839.65524.e0. PMID 15617591
- [Background] Kumar K, Buchser E, Linderoth B, Meglio M, Van Buyten JP. Avoiding complications from spinal cord stimulation: practical recommendations from an international panel of experts. Neuromodulation. 2007 Jan;10(1):24-33. doi: 10.1111/j.1525-1403.2007.00084.x. PMID 22151809
- [Background] Cruccu G, Aziz TZ, Garcia-Larrea L, Hansson P, Jensen TS, Lefaucheur JP, Simpson BA, Taylor RS. EFNS guidelines on neurostimulation therapy for neuropathic pain. Eur J Neurol. 2007 Sep;14(9):952-70. doi: 10.1111/j.1468-1331.2007.01916.x. PMID 17718686
- [Background] Schu S, Slotty PJ, Bara G, von Knop M, Edgar D, Vesper J. A prospective, randomised, double-blind, placebo-controlled study to examine the effectiveness of burst spinal cord stimulation patterns for the treatment of failed back surgery syndrome. Neuromodulation. 2014 Jul;17(5):443-50. doi: 10.1111/ner.12197. Epub 2014 Jun 19. PMID 24945621
- [Background] Meyerson BA, Linderoth B. Mechanisms of spinal cord stimulation in neuropathic pain. Neurol Res. 2000 Apr;22(3):285-92. doi: 10.1080/01616412.2000.11740672. PMID 10769822
- [Background] Wolter T. Spinal cord stimulation for neuropathic pain: current perspectives. J Pain Res. 2014 Nov 18;7:651-63. doi: 10.2147/JPR.S37589. eCollection 2014. PMID 25429237
- [Background] Kuechmann C, Valine T,Wolfe D. Could automatic position-adaptive stimulation be useful in spinal cord stimulation? Eur J Pain 2009;13:S243.
- [Background] De Ridder D, Vanneste S, Plazier M, van der Loo E, Menovsky T. Burst spinal cord stimulation: toward paresthesia-free pain suppression. Neurosurgery. 2010 May;66(5):986-90. doi: 10.1227/01.NEU.0000368153.44883.B3. PMID 20404705
- [Background] Al-Kaisy A, Van Buyten JP, Smet I, Palmisani S, Pang D, Smith T. Sustained effectiveness of 10 kHz high-frequency spinal cord stimulation for patients with chronic, low back pain: 24-month results of a prospective multicenter study. Pain Med. 2014 Mar;15(3):347-54. doi: 10.1111/pme.12294. Epub 2013 Dec 5. PMID 24308759
- [Background] Perruchoud C, Eldabe S, Batterham AM, Madzinga G, Brookes M, Durrer A, Rosato M, Bovet N, West S, Bovy M, Rutschmann B, Gulve A, Garner F, Buchser E. Analgesic efficacy of high-frequency spinal cord stimulation: a randomized double-blind placebo-controlled study. Neuromodulation. 2013 Jul-Aug;16(4):363-9; discussion 369. doi: 10.1111/ner.12027. Epub 2013 Feb 20. PMID 23425338